CLINICAL TRIAL: NCT01814046
Title: Phase II Study in Patients With Metastatic Ocular Melanoma Using a Non-Myeloablative Lymphocyte Depleting Regimen of Chemotherapy Followed by Infusion of Autologous Tumor-Infiltrating Lymphocytes With or Without High Dose Aldesleukin
Brief Title: Immunotherapy Using Tumor Infiltrating Lymphocytes for Patients With Metastatic Ocular Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Investigator left the National Institutes of Health (NIH)
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Steven Rosenberg, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 130093; 13-C-0093
Record Dates: First submitted 2013-03-15; First posted 2013-03-19 (Estimated); Results first posted 2017-07-24 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-09

CONDITIONS: Metastatic Ocular Melanoma; Metastatic Uveal Melanoma
Keywords: Metastatic; Ocular Melanoma; Autologous Tumor-Infiltrating Lymphocytes; Uveal Melanoma; Adoptive Cell Therapy
MeSH Terms: conditions — Uveal Melanoma; Neoplasm Metastasis | interventions — aldesleukin; Interleukin-2; Cyclophosphamide; fludarabine; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- cells + high dose aldesleukin (Experimental): Patients receiving cells + high dose aldesleukin
  Interventions: Drug: Aldesleukin; Drug: Cyclophosphamide; Drug: Fludarabine; Biological: Young Tumor Infiltrating Lymphocytes (TIL)
- cells and no high dose aldesleukin (Experimental): Patients receiving cells and no high dose aldesleukin
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: Young Tumor Infiltrating Lymphocytes (TIL)

INTERVENTIONS:
Drug: Aldesleukin — Aldesleukin 720,000 IU/kg intravenous (IV) (based on total body weight) over 15 minutes every eight hours (+/- 1 hour) beginning within 24 hours of cell infusion and continuing for up to 5 days (maximum of 15 doses) (only for cohort A).
  Other Names: Interleukin-2
  Arms: cells + high dose aldesleukin
Drug: Cyclophosphamide — Cyclophosphamide 60 mg/kg/day X 2 days intravenous (IV) in 250 ml dextrose 5% water (D5W) with Mesna 15 mg/kg/day X 2 days over 1 hr.
  Other Names: Cytoxan
Drug: Fludarabine — Fludarabine 25 mg/m^2/day intravenous piggy back (IVPB) daily over 30 minutes for 5 days.
  Other Names: Fludara
Biological: Young Tumor Infiltrating Lymphocytes (TIL) — Patients will receive non-myeloablative lymphodepleting preparative regimen consisting of cyclophosphamide and fludarabine followed by the administration of young TIL and high dose aldesleukin (Cohort A) or no aldesleukin (Cohort B). On day 0,cells (1x10e9 to 2x10e11) will be infused intravenously on the Patient Care Unit over 20-30 minutes.

SUMMARY:
Background:

- The National Cancer Institute (NCI) Surgery Branch has developed an experimental therapy that involves taking white blood cells from patients' tumors, growing them in the laboratory in large numbers, and then giving the cells back to the patient. These cells are called Tumor Infiltrating Lymphocytes, or TIL and we have given this type of treatment to over 200 patients with melanoma. This study will use chemotherapy to prepare the immune system before this white blood cell treatment. After receiving the cells, the drug aldesleukin (IL-2) may be given to help the cells stay alive longer.

Objectives:

- To see if chemotherapy and white blood cell therapy is a safe and effective treatment for advanced ocular melanoma.

Eligibility:

- Individuals at least greater than or equal to 16 years to less than or equal to 75 years who have advanced ocular melanoma.

Design:

* Work up stage: Patients will be seen as an outpatient at the National Institutes of Health (NIH) clinical Center and undergo a history and physical examination, scans, x-rays, lab tests, and other tests as needed.
* Surgery: If the patients meet all of the requirements for the study they will undergo surgery to remove a tumor that can be used to grow the TIL product.
* Leukapheresis: Patients may undergo leukapheresis to obtain additional white blood cells. {Leukapheresis is a common procedure, which removes only the white blood cells from the patient.}
* Treatment: Once their cells have grown, the patients will be admitted to the hospital for the conditioning chemotherapy, the TIL cells and aldesleukin. They will stay in the hospital for about 4 weeks for the treatment.
* Follow up: Patients will return to the clinic for a physical exam, review of side effects, lab tests, and scans about every 1-3 months for the first year, and then every 6 months to 1 year as long as their tumors are shrinking. Follow up visits take up to 2 days.

DETAILED DESCRIPTION:
Background:

* Metastatic ocular melanoma (OM) carries a poor prognosis with estimated survival of 4-6 months. There are no known effective systemic therapies. Metastatic OM is classified as an orphan disease and there are currently few clinical trial options for these patients. Thus, novel systemic approaches are desperately needed.
* Administration of autologous tumor infiltrating lymphocytes (TIL) generated from resected metastatic cutaneous melanoma can induce objective long-term tumor responses.
* Minimally invasive, safe, and effective surgical approaches have been developed in the Surgery Branch to procure liver tumor tissue for TIL generation.

Objectives:

* To determine whether autologous Young TIL infused with or without the administration of high-dose aldesleukin may result in clinical tumor regression in patients with metastatic ocular melanoma receiving a non-myeloablative lymphoid depleting preparative regimen.
* To study immunologic correlates associated with Young TIL therapy for ocular melanoma.
* To determine the toxicity of this treatment regimen.

Eligibility:

* Patients with metastatic ocular melanoma who are greater than or equal to 16 years of age, and are physically able to tolerate non-myeloablative chemotherapy. Patients who can tolerate high-dose aldesleukin will receive it following cell infusion; those who cannot tolerate high-dose aldesleukin due to medical comorbidities or refuse high dose aldesleukin will receive cell infusion without aldesleukin.
* There is no requirement for prior systemic therapies, given the lack of known effective systemic treatments for metastatic OM.

Design:

* Patients will undergo biopsy or resection to obtain tumor for generation of autologous TIL cultures and autologous cancer cell lines.
* All patients will receive a non-myeloablative lymphocyte depleting preparative regimen of cyclophosphamide and fludarabine.
* On day 0 patients will receive between 1x10^9 to 2x10^11 young TIL and then begin high dose aldesleukin (720,000 IU/kg intravenous (IV) every 8 hours for up to 15 doses) or no aldesleukin if they are not medically eligible to receive it.
* A complete evaluation of evaluable lesions will be conducted 4-6 weeks after the last dose of aldesleukin in the aldesleukin arm and 4-6 weeks after the cell administration in the no aldesleukin arm.
* Patients will be enrolled into two cohorts. The cohort receiving high-dose aldesleukin (cohort A) will be conducted using a small optimal two-stage Phase II design, initially 19 patients will be enrolled, and if 4 or more of the first 19 patients have a clinical response (partial response (PR) or complete response (CR), accrual will continue to 33 patients, targeting a 35% goal for objective response. For the cohort that will not receive aldesleukin (cohort B), the study will be conducted as a Minimax two-stage phase II trial. Initially 12 evaluable patients will be enrolled to this cohort, and if 1 or more the first 12 have a response, then accrual would continue until a total of 21 patients, targeting a 20% goal for objective response.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Measurable metastatic ocular melanoma.
  2. Confirmation of diagnosis of metastatic ocular melanoma by the Laboratory of Pathology of the National Cancer Institute (NCI).
  3. Patients with 3 or fewer brain metastases that are less than 1 cm in diameter and asymptomatic are eligible. Lesions that have been treated with stereotactic radiosurgery must be clinically stable for 1 month after treatment for the patient to be eligible. Patients with surgically resected brain metastases are eligible.
  4. Greater than or equal to 16 years of age and less than or equal to age 75.
  5. Able to understand and sign the Informed Consent Document
  6. Willing to sign a durable power of attorney
  7. Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0 or 1
  8. Life expectancy of greater than three months
  9. Patients of both genders must be willing to practice birth control from the time of enrollment on this study and for up to four months after receiving the treatment.
  10. Serology:

      * Seronegative for human immunodeficiency virus (HIV) antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune-competence and thus be less responsive to the experimental treatment and more susceptible to its toxicities.)
      * Seronegative for hepatitis B antigen, and seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, then patient must be tested for the presence of antigen by reverse transcription-polymerase chain reaction (RT-PCR) and be hepatitis C virus (HCV) ribonucleic acid (RNA) negative.
  11. Women of child-bearing potential must have a negative pregnancy test because of the potentially dangerous effects of the treatment on the fetus.
  12. Hematology

      * Absolute neutrophil count greater than 1000/mm^3 without the support of filgrastim
      * White blood cell (WBC) greater than or equal to 3000/mm^3
      * Platelet count greater than or equal 100,000/mm^3
      * Hemoglobin > 8.0 g/dl
  13. Chemistry:

      * Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) less than or equal to 3.5 times the upper limit of normal
      * Serum creatinine less than or equal to 1.6 mg/dl
      * Total bilirubin less than or equal to 2.0 mg/dl, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dl.
  14. More than four weeks must have elapsed since any prior systemic therapy at the time the patient receives the preparative regimen, and patients toxicities must have recovered to a grade 1 or less (except for toxicities such as alopecia or vitiligo).

Note: Patients may have undergone minor surgical procedures within the past 3 weeks, as long as all toxicities have recovered to grade 1 or less or as specified in the eligibility criteria.

EXCLUSION CRITERIA:

1. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the treatment on the fetus or infant.
2. Active systemic infections, coagulation disorders or other active major medical illnesses of the cardiovascular, respiratory or immune system, as evidenced by a positive stress thallium or comparable test, myocardial infarction, cardiac arrhythmias, obstructive or restrictive pulmonary disease.
3. Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
4. Concurrent opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities).
5. Concurrent systemic steroid therapy.
6. History of severe immediate hypersensitivity reaction to any of the agents used in this study.
7. The following patients will be excluded from the high-dose aldesleukin arm (but may be eligible for cells alone arm):

   1. History of coronary revascularization or ischemic symptoms
   2. Documented left ventricular ejection fraction (LVEF) of less than or equal to 45%. Testing is required in patients with:

      * Clinically significant atrial and/or ventricular arrhythmias including but not limited to: atrial fibrillation, ventricular tachycardia, second or third degree heart block
      * Age greater than or equal to 60 years old
   3. Clinically significant patient history which in the judgment of the Principal Investigator would compromise the patients ability to tolerate aldesleukin

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-03-01 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Rosenberg, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Woodman SE. Metastatic uveal melanoma: biology and emerging treatments. Cancer J. 2012 Mar-Apr;18(2):148-52. doi: 10.1097/PPO.0b013e31824bd256. PMID 22453016
- [Background] Rosenberg SA, Yang JC, Sherry RM, Kammula US, Hughes MS, Phan GQ, Citrin DE, Restifo NP, Robbins PF, Wunderlich JR, Morton KE, Laurencot CM, Steinberg SM, White DE, Dudley ME. Durable complete responses in heavily pretreated patients with metastatic melanoma using T-cell transfer immunotherapy. Clin Cancer Res. 2011 Jul 1;17(13):4550-7. doi: 10.1158/1078-0432.CCR-11-0116. Epub 2011 Apr 15. PMID 21498393
- [Background] Singh AD, Turell ME, Topham AK. Uveal melanoma: trends in incidence, treatment, and survival. Ophthalmology. 2011 Sep;118(9):1881-5. doi: 10.1016/j.ophtha.2011.01.040. Epub 2011 Jun 24. PMID 21704381
- [Derived] Chandran SS, Somerville RPT, Yang JC, Sherry RM, Klebanoff CA, Goff SL, Wunderlich JR, Danforth DN, Zlott D, Paria BC, Sabesan AC, Srivastava AK, Xi L, Pham TH, Raffeld M, White DE, Toomey MA, Rosenberg SA, Kammula US. Treatment of metastatic uveal melanoma with adoptive transfer of tumour-infiltrating lymphocytes: a single-centre, two-stage, single-arm, phase 2 study. Lancet Oncol. 2017 Jun;18(6):792-802. doi: 10.1016/S1470-2045(17)30251-6. Epub 2017 Apr 7. PMID 28395880
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-C-0093.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients experiencing a sustained stable disease, partial or complete response may receive a second treatment when progression by the Response Evaluation Criteria in Solid Tumors (RECIST) criteria is documented after evaluation by the principal investigator. Retreatment will consist of the same regimen that they had been given safely previously.
Groups:
- Cells and no High Dose Aldesleukin: Patients receiving cells and no high dose aldesleukin
  Cyclophosphamide: Cyclophosphamide 60 mg/kg/day X 2 days intravenous (IV) in 250 ml dextrose 5% water (D5W) with Mesna 15 mg/kg/day X 2 days over 1 hr.
  Fludarabine: Fludarabine 25 mg/m^2/day intravenous piggy back (IVPB) daily over 30 minutes for 5 days.
  Young TIL: Patients will receive non-myeloablative lymphodepleting preparative regimen consisting of cyclophosphamide and fludarabine followed by the administration of young TIL and high dose aldesleukin (Cohort A) or no aldesleukin (Cohort B). On day 0,cells (1x10e9 to 2x10e11) will be infused intravenously on the Patient Care Unit over 20-30 minutes.
- Cells + High-Dose Aldesleukin Retreatment: Patients experiencing a sustained stable disease, partial or complete response may receive a second treatment when progression by the Response Evaluation Criteria in Solid Tumors (RECIST) criteria is documented after evaluation by the principal investigator. Retreatment will consist of the same regimen that they had been given safely previously.
Period: Drug Administration
Arm/Group | Cells + High Dose Aldesleukin | Cells and no High Dose Aldesleukin | Cells + High-Dose Aldesleukin Retreatment
Started | 22 | 2 | 0
Completed | 21 | 2 | 0
Not Completed | 1 | 0 | 0
Not completed — Death due to complications of RSV | 1 | 0 | 0
Period: Retreatment
Arm/Group | Cells + High Dose Aldesleukin | Cells and no High Dose Aldesleukin | Cells + High-Dose Aldesleukin Retreatment
Started | 0 | 0 | 3
Completed | 0 | 0 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cells + High Dose Aldesleukin | Cells and no High Dose Aldesleukin | Total
Number analyzed (Participants) | 22 | 2 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 1 | 23
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (8.4) | 64 (4.2) | 57.85 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 0 | 8
  Male | 14 | 2 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 22 | 2 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 22 | 2 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 2 | 24

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Ocular Melanoma Treated With Young Tumor Infiltrating Lymphocytes (TIL) With or Without High Dose Aldesleukin With an Objective Response Rate of (Complete Response (CR) + Partial Response (PR))
Description: Objective response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST). Complete response is disappearance of all target lesions. Partial response is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline sum LD.
Time Frame: approximately 3 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cells + High Dose Aldesleukin | Cells and no High Dose Aldesleukin
Number analyzed (Participants) | 22 | 2
percentage of participants
  Complete Response (CR) | 4.54 [0 to 22.8] | 0 [0 to 0]
  Partial Response (PR) | 31.81 [13.9 to 54.9] | 0 [0 to 0]

2. Secondary Outcome: Count of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria in Adverse Events (CTCAE v3.0)
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v3.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: 46 months and 12 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cells + High Dose Aldesleukin | Cells and no High Dose Aldesleukin
Number analyzed (Participants) | 22 | 2
Participants | 22 | 2

3. Other Pre Specified Outcome: Count of Participants With Changes in Visual Symptoms
Description: Visual symptoms (e.g., blurred) were evaluated and if changes had occurred from baseline, i.e. in visual acuity, an ophthalmologic consult was performed.
Time Frame: 6 weeks (+/- 2 weeks)
Population: One out of 24 subjects had blurred vision.
Measure: Count of Participants; unit: Participants
Arm/Group | Cells + High Dose Aldesleukin | Cells and no High Dose Aldesleukin
Number analyzed (Participants) | 22 | 2
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: 46 months and 12 days
Groups:
- Cells + High-Dose Aldesleukin: Patients receiving cells + high dose aldesleukin
  Aldesleukin: Aldesleukin 720,000 IU/kg intravenous (IV) (based on total body weight) over 15 minutes every eight hours (+/- 1 hour) beginning within 24 hours of cell infusion and continuing for up to 5 days (maximum of 15 doses) (only for cohort A).
  Cyclophosphamide: Cyclophosphamide 60 mg/kg/day X 2 days intravenous (IV) in 250 ml dextrose 5% water (D5W) with Mesna 15 mg/kg/day X 2 days over 1 hr.
  Fludarabine: Fludarabine 25 mg/m^2/day intravenous piggy back (IVPB) daily over 30 minutes for 5 days.
  Young tumor infiltrating lymphocytes (TIL): Patients will receive non-myeloablative lymphodepleting preparative regimen consisting of cyclophosphamide and fludarabine followed by the administration of young TIL and high dose aldesleukin (Cohort A) or no aldesleukin (Cohort B). On day 0,cells (1x10e9 to 2x10e11) will be infused intravenously on the Patient Care Unit over 20-30 minutes.
- Cells and No High-Dose Aldesleukin: Patients receiving cells and no high dose aldesleukin
  Cyclophosphamide: Cyclophosphamide 60 mg/kg/day X 2 days intravenous (IV) in 250 ml dextrose 5% water (D5W) with Mesna 15 mg/kg/day X 2 days over 1 hr.
  Fludarabine: Fludarabine 25 mg/m^2/day intravenous piggy back (IVPB) daily over 30 minutes for 5 days.
  Young TIL: Patients will receive non-myeloablative lymphodepleting preparative regimen consisting of cyclophosphamide and fludarabine followed by the administration of young TIL and high dose aldesleukin (Cohort A) or no aldesleukin (Cohort B). On day 0,cells (1x10e9 to 2x10e11) will be infused intravenously on the Patient Care Unit over 20-30 minutes.
Arm/Group | Cells + High-Dose Aldesleukin | Cells and No High-Dose Aldesleukin | Cells + High-Dose Aldesleukin Retreatment
All-Cause Mortality (participants affected / at risk) | 1/22 | 0/2 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/22 | 0/2 | 2/3
Other Adverse Events (participants affected / at risk) | 22/22 | 2/2 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cells + High-Dose Aldesleukin (N=22) | Cells and No High-Dose Aldesleukin (N=2) | Cells + High-Dose Aldesleukin Retreatment (N=3)
CNS cerebrovascular ischemia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Death not associated with CTCAE term::Multi-organ failure (General disorders) | 1 (1) | 0 (0) | 0 (0)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — (ANC <1.0 x 10e9/L)::Blood
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Neuropathy: motor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Platelets (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cells + High-Dose Aldesleukin (N=22) | Cells and No High-Dose Aldesleukin (N=2) | Cells + High-Dose Aldesleukin Retreatment (N=3)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 0 (0)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Alkaline phosphatase (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 1 (1)
Cardiac Arrhythmia - Other (Specify, cardiac arrhythmia) (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Creatinine (Metabolism and nutrition disorders) | 7 (7) | 0 (0) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0) | 0 (0)
Edema: viscera (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 5 (5) | 0 (0) | 2 (2)
Febrile neutropenia (Infections and infestations) | 6 (6) | 1 (1) | 0 (0) — (fever of unknown origin without clinically or microbiologically documented infection) (ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Hemoglobin (Blood and lymphatic system disorders) | 14 (14) | 0 (0) | 2 (2)
Hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Infections and infestations) | 6 (7) | 0 (0) | 1 (1) — (ANC <1.0 x 10e9/L)::Blood
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 12 (12) | 1 (1) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 22 (23) | 2 (2) | 3 (3)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 22 (22) | 2 (2) | 1 (1)
PTT (Partial Thromboplastin Time) (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (2)
Platelets (Blood and lymphatic system disorders) | 22 (22) | 2 (2) | 2 (2)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal/Genitourinary - Other (Specify, decrease urine output) (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal/Genitourinary - Other (Specify, oliguriat) (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Supraventricular and nodal arrhythmia::Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Vision-blurred vision (Eye disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2017-05-05): https://cdn.clinicaltrials.gov/large-docs/46/NCT01814046/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-06-30): https://cdn.clinicaltrials.gov/large-docs/46/NCT01814046/Prot_SAP_001.pdf